CLINICAL TRIAL: NCT01727284
Title: Technical Success, Safety, and Short and Long-term Efficacy for MR-Guided Cryoablation of Prostate Bed Recurrences
Brief Title: MR-Guided Cryoablation of Prostate Bed Recurrences
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, Assistant Professor of Radiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-002245; NCI-2023-01699 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Prostate Tumors
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR-guided cryoablation (freezing of tissue and/or tumors) (Experimental): Patients undergo cryoablation using the Galil MR-compatible cryoablation system and MRI while on study.
  Interventions: Procedure: MR-guided cryoablation

INTERVENTIONS:
Procedure: MR-guided cryoablation

SUMMARY:
The purpose of this research is to see if MR-guided cryoablation can effectively treat prostate tumor recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with "biopsy proven" soft tissue tumor recurrences of prostate fossa
* Surgery is not a desirable alternative therapy at the time of enrollment
* Radiation therapy has failed or not indicated or can be safely postponed
* Tumor size is < 5 cm at its largest diameter
* Tumor does not encompass the rectal wall or external urethral sphincter
* Patient is able to undergo MRI

Exclusion Criteria:

* N/A

Ages: 30 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of target lesion at 3-6, 12, 24, and 36 month imaging follow-up | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials